CLINICAL TRIAL: NCT06948721
Title: Study of the Participation of People With Aphasia Post Stroke and Their Caregivers in Valladolid Region (Spain)
Acronym: SPART-A
Status: Not yet recruiting | Type: Observational
Sponsor: Centro Integral de Rehabilitación (Other)
Responsible Party: Principal Investigator, Jorge Alegre Ayala, Principal Investigator, Centro Integral de Rehabilitación
Other Study IDs: CIRON
Record Dates: First submitted 2025-04-11; First posted 2025-04-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Aphasia
Keywords: Aphasia post stroke; caregiver; community participation; occupational therapy; Speech Language Therapy
MeSH Terms: conditions — Stroke; Aphasia; Communication Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- people with aphasia post stroke
- Caregivers of people with aphasia post stroke

SUMMARY:
The objective of this study is to determine the level of community participation of people with post-stroke aphasia and their caregivers, as well as the factors that facilitate or interfere with this participation in the Valladolid region (Spain).

The main questions that this study aims to answer are:

1. What is the retained activities of the people with aphasia post-stroke?
2. What is the retained activities of the caregivers of people with aphasia post-stroke?
3. What factors influence the community participation of people with aphasia post-stroke and their caregivers?

ELIGIBILITY:
Inclusion Criteria:

* Chronic Stroke (stroke onset above six months).
* Aphasia post stroke.
* Residents in Valladolid Region.
* Age over 18 years.
* Ability to walk equal to or greater than 3 according to the Functional Ambulation Category (FAC).
* Informed consent acceptance.

Exclusion Criteria:

* Stroke onset below of Six months
* Age under 18 years
* Both in the case of the person with aphasia and their caregiver, presence of other pathologies that affect functional independence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants in the study (people with aphasia and their caregivers) will be drawn from the registry of people treated at the companies CIRONBRAIN and CIRONLAB, which comprise the research team. Sample recruitment will also be conducted through CIRONBRAIN's social media channels, and through requests for collaboration with local disability organizations and healthcare professionals in the Valladolid region who are familiar with the project and who may be eligible for selection.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-06 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Activity Card Sort | Baseline
  The Activity Card Sort will determine the level of participation maintained by people with aphasia and their caregivers at the time of the assessment. It will provide data on overall participation, as well as participation in leisure, social, educational, and work activities. The Activity Card Sort scale scores range from 0 to 100%. Higher percentages, better.

SECONDARY OUTCOMES:
The Western Aphasia Battery (WAB) | Baseline
  The Western Aphasia Battery (WAB) is a tool used to assess the linguistic skills (information content, fluency, auditory comprehension, repetition, naming and word finding, reading, and writing) and nonlinguistic skills (drawing, block design, calculation, and praxis) of adults with aphasia. This provides information for the diagnosis of the type of aphasia. The Western Aphasia Battery uses an Aphasia Quotient (AQ) to assess the severity of aphasia, with scores ranging from 0 to 100. Higher score, less severity of aphasia.
Barthel Index (BI) | Baseline
  The BI assesses the level of functional independence in basic activities of daily living (eating, hygiene, dressing, mobility, etc.). Barthel index scores range from 0 to 100 points. Higher scores, better.
Zarit Caregiver Burden Interview (ZBI) | Baseline
  The aim of the Zarit Caregiver Burden Interview (ZBI) is to assess the perceived burden experienced by caregivers, particularly in terms of the physical, emotional, social, and financial impacts of caregiving. The Zarit Caregiver Burden Interview scale scores range from 22 to 110 points. Higher scores indicate worse outcomes.
Six-Minute Walk Test (6MWT) | Baseline
  The Six-Minute Walk test aims to assess a person's functional exercise capacity by measuring the distance they can walk in six minutes on a flat surface. Higher score, better.
Ten-Meter Walk Test (10MWT) | Baseline.
  The Ten-Meter Walk Test evaluates walking speed over a short distance (10 meters). This scale provides data on normal speed and fast speed. Higher speed, better.
Hospital Anxiety and Depression Scale | Baseline
  The purpose of the Hospital Anxiety and Depression Scale is identify depression and anxiety among physically ill patients, through a brief questionnaire which involves both dimensions. The scoring of the Hospital Anxiety and Depression Scale 0-21 for each subscale, with higher scores indicating greater anxiety or depression.

IPD SHARING:
Plan to Share IPD: No